CLINICAL TRIAL: NCT01634555
Title: A Study to Evaluate the Potential of Concomitant Ramucirumab to Affect the Pharmacokinetics of Irinotecan and Its Metabolite SN-38 When Coadministered With Folinic Acid and 5 Fluorouracil in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study to Assess the Pharmacokinetics of Ramucirumab (IMC-1121B) in Combination With FOLFIRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14433; CP12-1033 (Other: ImClone Systems); I4T-IE-JVCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumors
Keywords: Advanced Malignant Solid Tumors
MeSH Terms: interventions — Ramucirumab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ramucirumab (IMC-1121B) and FOLFIRI (Experimental): Treatment is sequential, Ramucirumab (IMC-1121B) will be administered before FOLFIRI ((Irinotecan + Folinic acid + 5-Fluorouracil). FOLFIRI will be administered each cycle and Ramucirumab (IMC-1121B) will be administered beginning from Cycle 2 (2-week cycle).
  Interventions: Biological: Ramucirumab (IMC-1121B); Drug: Irinotecan; Drug: Folinic acid; Drug: 5-Fluorouracil

INTERVENTIONS:
Biological: Ramucirumab (IMC-1121B) — Ramucirumab (IMC-1121B) 8 milligrams per kilogram (mg/kg), administered as an intravenous (IV) infusion on Day 1 of each 2-week cycle (except Cycle 1)
  Other Names: IMC-1121B; LY3009806
Drug: Irinotecan — 180 milligrams per square meter (mg/m²) administered IV on Day 1 of each cycle
Drug: Folinic acid — 400 mg/m² administered IV on Day 1 of each cycle
Drug: 5-Fluorouracil — 400 mg/m² bolus over 2 to 4 minutes administered IV on Day 1 of each cycle, followed by 2400 mg/m² administered IV over 46 to 48 hours on Days 1 and 2 of each cycle

SUMMARY:
The purpose of this study is to assess the effect of concomitant ramucirumab (IMC-1121B) on the pharmacokinetics of irinotecan and its metabolite SN-38 when coadministered with folinic acid and 5-fluorouracil, in participants with advanced malignant solid tumors resistant to standard therapy or for which no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

* Has histologic or cytologic documentation of a malignant solid tumor
* Has an advanced solid tumor that is resistant to standard therapy or for which no standard therapy is available
* Has resolution to Grade ≤1, per the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v. 4.0), of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Has adequate hematologic, coagulation, and hepatic function
* Has serum creatinine ≤ 1.5 x upper limit of normal (ULN)
* Urinary protein is <2+ on dipstick or routine urinalysis (UA) at study entry
* Women with childbearing potential must have a negative serum or urine pregnancy test
* Eligible participants of reproductive potential (both sexes) agree to use adequate method of contraception during the study period and for 12 weeks after the last dose of study medication

Exclusion Criteria:

* Has received a therapeutic monoclonal antibody within the last 42 days
* Has received cytotoxic chemotherapy within the last 21 days
* Has received radiotherapy within the last 14 days
* Are currently enrolled in, or discontinued within the last 14 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Has a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism during the last 3 months
* Has an uncontrolled illness, including, but not limited to uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness/social situations, or any other serious uncontrolled medical disorders
* Has experienced any arterial thromboembolic event within the last 6 months
* Has known leptomeningeal disease or brain metastases or uncontrolled spinal cord compression
* Has an ongoing or active infection requiring parenteral antibiotic, antifungal, or antiviral therapy
* Has known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness
* Has received a prior organ or transplantation
* Has undergone major surgery within the last 28 days
* Has had a serious nonhealing wound, ulcer, or bone fracture within the last 28 days
* Has an elective or planned major surgery to be performed during the course of the trial
* Has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection, Crohn's disease, ulcerative colitis, or chronic diarrhea
* Has experienced a Grade 3 or higher bleeding event within the last 3 months
* Has a known history or clinical evidence of Gilbert's Syndrome, or is known to have any of the following genotypes: uridine diphosphate glucuronosyltransferase isoform 1A1 (UGT1A1)*6/*6, UGT1A1*28/*28, or UGT1A1*6/*28
* Has received clinically relevant inhibitors or inducers of cytochrome P (CYP) 450 CYP3A4/5 or CYP2C9 and/or isoenzymes within the last 3 weeks
* Has cirrhosis at a level of Child-Pugh B (or worse), or cirrhosis and a history of hepatic encephalopathy, or ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramucirumab (IMC-1121B) and FOLFIRI: Treatment is sequential. Ramucirumab (IMC-1121B) was administered before FOLFIRI (Irinotecan + Folinic acid + 5-Fluorouracil) during Cycles 2+
  Ramucirumab (IMC-1121B): 8 milligrams per kilogram (mg/kg) administered as an intravenous (IV) infusion on Day 1 of each 2-week cycle (except Cycle 1)
  Irinotecan: 180 milligrams per square meter (mg/m²) administered IV on Day 1 of each 2-week cycle
  Folinic acid: 400 mg/m² administered IV on Day 1 of each 2-week cycle
  5-Fluorouracil: 400 mg/m² bolus over 2 to 4 minutes administered IV on Day 1 of each cycle, followed by 2400 mg/m² administered IV over 46 to 48 hours on Days 1 and 2 of each 2-week cycle
Period: Overall Study
Arm/Group | Ramucirumab (IMC-1121B) and FOLFIRI
Started | 29
Received at Least 1 Dose of Study Drug | 29
Drug-Drug Interaction (DDI) Population | 25 (Completed the required treatment in Cycle 1, Day 1 and Cycle 2, Day 1.)
Completed | 25 (Completed the required treatment and assessment.)
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Ramucirumab (IMC-1121B) and FOLFIRI: Treatment is sequential. Ramucirumab (IMC-1121B) was administered before FOLFIRI (Irinotecan + Folinic acid + 5-Fluorouracil) during Cycles 2+
  Ramucirumab (IMC-1121B): 8 mg/kg administered as IV infusion on Day 1 of each 2-week cycle (except Cycle 1)
  Irinotecan: 180 mg/m² administered IV on Day 1 of each 2-week cycle
  Folinic acid: 400 mg/m² administered IV on Day 1 of each 2-week cycle
  5-Fluorouracil: 400 mg/m² bolus over 2 to 4 minutes administered IV on Day 1 of each 2-week cycle, followed by 2400 mg/m² administered IV over 46 to 48 hours on Days 1 and 2 of each cycle
Arm/Group | Ramucirumab (IMC-1121B) and FOLFIRI
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Dose-Normalized Area Under the Concentration Versus Time Curve of Irinotecan and Its Metabolite SN-38 From Time Zero to Infinity [AUC(0-∞)] in Cycle 1
Description: Dose-normalized AUC(0-∞) was calculated from AUC(0-∞) divided by the dose. Data presented are Geometric Least Squares (Geo LS) means. Geo LS means were adjusted for cycle, participant and random error.
Time Frame: Cycle 1: 0, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 22, 25, 28, 31, 34, 48, 72, 96 and 168 hours post-irinotecan infusion
Population: All participants in DDI population (who completed the required treatment in Cycle 1, Day 1 and Cycle 2, Day 1) and had sufficient concentration data to calculate irinotecan and its metabolite SN-38 AUC(0-∞) in Cycle 1.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms*hour/milliliter/milligram
Groups:
- FOLFIRI (Cycle 1): Irinotecan: 180 mg/m² administered IV on Day 1 of Cycle 1 (2-week cycle)
  Folinic acid: 400 mg/m² administered IV on Day 1 of Cycle 1 (2-week cycle)
  5-Fluorouracil: 400 mg/m² bolus over 2 to 4 minutes administered IV on Day 1, followed by 2400 mg/m² administered IV over 46 to 48 hours on Days 1 and 2 of Cycle 1 (2-week cycle)
Arm/Group | FOLFIRI (Cycle 1)
Number analyzed (Participants) | 25
nanograms*hour/milliliter/milligram
  Irinotecan | 22.12 [19.72 to 24.82]
  Metabolite SN-38 | 0.81 [0.70 to 0.93]

2. Primary Outcome: Pharmacokinetics: Dose-Normalized AUC(0-∞) of Irinotecan and Its Metabolite SN-38 in Cycle 2
Description: Dose-normalized AUC(0-∞) was calculated from AUC(0-∞) divided by the dose. Data presented are Geo LS means. Geo LS means were adjusted for cycle, participant and random error.
Time Frame: Cycle 2: 0, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 22, 25, 28, 31, 34, 48, 72, 96 and 168 hours post-irinotecan infusion
Population: All participants in DDI population (who completed the required treatment in Cycle 1, Day 1 and Cycle 2, Day 1) and had sufficient concentration data to calculate irinotecan and its metabolite SN-38 AUC(0-∞) in Cycle 2.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms*hour/milliliter/milligram
Groups:
- Ramucirumab + FOLFIRI (Cycle 2): Ramucirumab (IMC-1121B): 8 mg/kg administered as IV infusion on Day 1 of Cycle 2 (2-week cycle)
  Irinotecan: 180 mg/m² administered IV on Day 1 of both Cycles 1 and 2 (2-week cycle)
  Folinic acid: 400 mg/m² administered IV on Day 1 of both Cycles 1 and 2 (2-week cycle)
  5-Fluorouracil: 400 mg/m² bolus over 2 to 4 minutes administered IV on Day 1 of Cycles 1 and 2, followed by 2400 mg/m² administered IV over 46 to 48 hours on Days 1 and 2 of both Cycles 1 and 2 (2-week cycle)
Arm/Group | Ramucirumab + FOLFIRI (Cycle 2)
Number analyzed (Participants) | 25
nanograms*hour/milliliter/milligram
  Irinotecan | 20.56 [18.33 to 23.06]
  Metabolite SN-38: number analyzed (Participants) | 24
  Metabolite SN-38 | 0.77 [0.67 to 0.89]
Statistical Analysis 1: Comparison: Ramucirumab + FOLFIRI (Cycle 2); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geo LS mean is AUC(0-∞) of Cycle 2/Cycle 1 for Irinotecan; Ratio of Geo LS means = 0.93, 90% CI 2-sided [0.83 to 1.05]
Statistical Analysis 2: Comparison: Ramucirumab + FOLFIRI (Cycle 2); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geo LS mean is AUC(0-∞) of Cycle 2/Cycle 1 for Metabolite SN-38; Ratio of Geo LS means = 0.95, 90% CI 2-sided [0.88 to 1.04]

3. Primary Outcome: Pharmacokinetics: Dose-Normalized Maximum Observed Drug Concentration (Cmax) of Irinotecan and Its Metabolite SN-38 in Cycle 1
Description: Dose-normalized Cmax was calculated from Cmax divided by the dose. Data presented are Geo LS means. Geo LS means were adjusted for cycle, participant and random error.
Time Frame: Cycle 1: 0, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 22, 25, 28, 31, 34, 48, 72, 96 and 168 hours post-irinotecan infusion
Population: All participants in DDI population (who completed the required treatment in Cycle 1, Day 1 and Cycle 2, Day 1) and had sufficient concentration data to calculate irinotecan and its metabolite SN-38 Cmax in Cycle 1.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms/milliliter/milligram
Arm/Group | FOLFIRI (Cycle 1)
Number analyzed (Participants) | 23
nanograms/milliliter/milligram
  Irinotecan | 3.18 [2.91 to 3.48]
  Metabolite SN-38 | 0.05 [0.04 to 0.06]

4. Primary Outcome: Pharmacokinetics: Dose-Normalized Cmax of Irinotecan and Its Metabolite SN-38 in Cycle 2
Description: as for outcome 3
Time Frame: Cycle 2: 0, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 22, 25, 28, 31, 34, 48, 72, 96 and 168 hours post-irinotecan infusion
Population: All participants in DDI population (who completed the required treatment in Cycle 1, Day 1 and Cycle 2, Day 1) and had sufficient concentration data to calculate irinotecan and its metabolite SN-38 Cmax in Cycle 2.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms/milliliter/milligram
Arm/Group | Ramucirumab + FOLFIRI (Cycle 2)
Number analyzed (Participants) | 23
nanograms/milliliter/milligram
  Irinotecan | 3.31 [3.02 to 3.62]
  Metabolite SN-38 | 0.05 [0.04 to 0.06]
Statistical Analysis 1: Comparison: Ramucirumab + FOLFIRI (Cycle 2); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geo LS mean is Cmax of Cycle 2/Cycle 1 for Irinotecan; Ratio of Geo LS means = 1.04, 90% CI 2-sided [0.97 to 1.12]
Statistical Analysis 2: Comparison: Ramucirumab + FOLFIRI (Cycle 2); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geo LS mean is Cmax of Cycle 2/Cycle 1 for Metabolite SN-38; Ratio of Geo LS means = 0.97, 90% CI 2-sided [0.85 to 1.12]

5. Secondary Outcome: Pharmacokinetics: Cmax of Ramucirumab (IMC-1121B)
Time Frame: Cycle 2: -2, -1, -0.5, 0, 2, 3, 4, 5, 8, 10, 25, 48, 72, 96, 168, 264, 336 hours post-ramucirumab (IMC-1121B) infusion
Population: All participants who received study drug and had sufficient concentration data to calculate ramucirumab (IMC-1121B) Cmax in Cycle 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Ramucirumab + FOLFIRI (Cycle 2)
Number analyzed (Participants) | 25
micrograms/milliliter (µg/mL) | 201.6 (31)

6. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Drug Antibodies (TE-ADA)
Description: Number of participants with positive treatment emergent anti-ramucirumab antibodies was summarized by treatment group.
Time Frame: Up To 2 Years
Population: All participants with both baseline and at least one post baseline ADA assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + FOLFIRI (Cycle 2)
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: Up To 2 Years
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Ramucirumab (IMC-1121B) and FOLFIRI: Treatment is sequential. Ramucirumab (IMC-1121B) was administered before FOLFIRI (Irinotecan + Folinic acid + 5-Fluorouracil) during Cycles 2+
  Ramucirumab (IMC-1121B): 8 mg/kg, administered as IV infusion on Day 1 of each 2-week cycle (except Cycle 1)
  Irinotecan: 180 mg/m² administered IV on Day 1 of each 2-week cycle
  Folinic acid: 400 mg/m² administered IV on Day 1 of each 2-week cycle
  5-Fluorouracil: 400 mg/m² bolus over 2 to 4 minutes administered IV on Day 1 of each 2-week cycle, followed by 2400 mg/m² administered IV over 46 to 48 hours on Days 1 and 2 of each cycle
Arm/Group | Ramucirumab (IMC-1121B) and FOLFIRI
Serious Adverse Events (participants affected / at risk) | 11/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (IMC-1121B) and FOLFIRI (N=29)
Ascites (Gastrointestinal disorders) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (4)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ramucirumab (IMC-1121B) and FOLFIRI (N=29)
Anaemia (Blood and lymphatic system disorders) | 15 (48)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 7 (18)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 15 (28)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (14)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 15 (23)
Ascites (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (17)
Diarrhoea (Gastrointestinal disorders) | 20 (32)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 2 (4)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 17 (28)
Oral pain (Gastrointestinal disorders) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 2 (4)
Tongue discolouration (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (14)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 21 (45)
Mucosal inflammation (General disorders) | 11 (16)
Oedema peripheral (General disorders) | 7 (11)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (4)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 8 (18)
Blood alkaline phosphatase increased (Investigations) | 10 (13)
Blood creatinine increased (Investigations) | 2 (6)
Blood lactate dehydrogenase increased (Investigations) | 3 (3)
Haemoglobin decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 4 (7)
Weight decreased (Investigations) | 10 (15)
White blood cell count decreased (Investigations) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 15 (30)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (9)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 (24)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 5 (6)
Neuropathy peripheral (Nervous system disorders) | 6 (9)
Tremor (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (6)
Nocturia (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 7 (11)
Erectile dysfunction (Reproductive system and breast disorders) | 1/15 (3)
Testicular pain (Reproductive system and breast disorders) | 1/15 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (7)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (7)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.